CLINICAL TRIAL: NCT03621150
Title: Comparative Study Between Dynamic Ultrasound and MRI in Evaluation of Tendino-ligamentous Injuries Around the Ankle Joint
Brief Title: Dynamic Ultrasound in Evaluation of Tendo-ligamentous Ankle Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Shaker Abolela Shehata, Principal investigator, Assiut University
Other Study IDs: Dynamic ankle ultrasound
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Tendinoligamentous Injury of the Ankle
Keywords: mri; musculoskeletal ultrasound; tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients complaining of ankle pain, swelling or dysfunction underwent ultrasound examination and then MRI as a reference to compare the diagnostic accuracy of ultrasonography in the assessment of tendino-ligamentous injuries around the ankle joint

SUMMARY:
Several imaging modalities, such as computed tomography, magnetic resonance imaging, and ultrasound (US) can be used to evaluate the ankle. However, US has several benefits for the evaluation of the tendons and ligaments of the ankle, such as its suitability to be integrated with a dynamic assessment and a stress test, its ability to provide real-time analysis, its avoidance of the risk of radiation exposure, and its cost-effectiveness. US is especially powerful when used to evaluate a tear, subluxation, or dislocation in a dynamic examination and when performing a comparison with the contralateral extremity. Dynamic imaging with muscle contraction or passive movement is often helpful. Additionally, Doppler imaging may be used to distinguish small intrasubstance tears from blood vessels that can occur in a tendinopathic tendon.

DETAILED DESCRIPTION:
Ankle injuries account for approximately 14% of sports-related orthopedic emergency visits. Various pathological conditions can affect the ankle, including trauma, overuse disorders, and inflammatory conditions.

Several imaging modalities, such as computed tomography, magnetic resonance imaging, and ultrasound (US) can be used to evaluate the ankle. However, US has several benefits for the evaluation of the tendons and ligaments of the ankle, such as its suitability to be integrated with a dynamic assessment and a stress test, its ability to provide real-time analysis, its avoidance of the risk of radiation exposure, and its cost-effectiveness. US is especially powerful when used to evaluate a tear, subluxation, or dislocation in a dynamic examination and when performing a comparison with the contralateral extremity. Dynamic imaging with muscle contraction or passive movement is often helpful. Additionally, Doppler imaging may be used to distinguish small intrasubstance tears from blood vessels that can occur in a tendinopathic tendon.

Approximately 85%of them are due to inversion forces and, therefore, involve the lateral collateral ligamentous complex. A Grade I sprain is a mild injury limited to microtears and stretching of the ligaments. Grade II sprains are partial macroscopic tears and in Grade III sprains the ligament has ruptured completely. There is general agreement that the overwhelming majority of Grade I and II sprains heal uneventfully with conservative care. Treatment of Grade III sprains is more controversial: some practitioners prefer operative repair, at least for high-performance athletes and others prefer a regimen of casting and physical therapy, which is the case in our institution. The proper role of imaging in the diagnosis of ankle sprains includes first of all conventional radiographs to ensure a fracture is not overlooked. Ultrasound is will be used to evaluate disorders of the musculoskeletal system, and because of their size and superficial location the ankle tendons can be well evaluated

ELIGIBILITY:
Inclusion Criteria:

* patients complaining of unilateral ankle joint pain (acute or chronic).

Exclusion Criteria:

* previous ankle surgery, interventional Intra-articular procedures (previous arthroscope, injections),
* Systemic inflammatory disorders (collagen diseases),
* Diagnosed osseous lesions.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: no gender based Age 15-60 -y-old Complaining from unilateral ankle pain or instability
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of ankle tendi-ligamentous injury by dynamic ultrasound and MRI | 1 month
  Approximately 85%of anke tendo-ligamentous injuries are due to inversion forces and, therefore involve the lateral collateral ligamentous complex.
  * Grade I sprain is a mild injury limited to microtears and stretching of the ligaments.
  * Grade II sprains are partial macroscopic tears
  * Grade III sprains the ligament has ruptured completely.

REFERENCES:
- [Background] Bianchi S, Martinoli C, Gaignot C, De Gautard R, Meyer JM. Ultrasound of the ankle: anatomy of the tendons, bursae, and ligaments. Semin Musculoskelet Radiol. 2005 Sep;9(3):243-59. doi: 10.1055/s-2005-921943. PMID 16247724
- [Background] Khoury V, Guillin R, Dhanju J, Cardinal E. Ultrasound of ankle and foot: overuse and sports injuries. Semin Musculoskelet Radiol. 2007 Jun;11(2):149-61. doi: 10.1055/s-2007-1001880. PMID 18095247